CLINICAL TRIAL: NCT00806143
Title: Bilateral Versus Monolateral Repetitive Transcranial Stimulation in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Neuroscience, Florence, Italy (Other)
Responsible Party: Stefano Pallanti, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMSDEP
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Major Depression
Keywords: Depression; TMS
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): patients will undergo sequential bilateral rTMS treatment
  Interventions: Device: repetitive transcranial stimulation (rTMS)
- 2 (Active Comparator): patients will undergo unilateral low frequency right sided DLPFC rTMS
  Interventions: Device: unilateral stimulation

INTERVENTIONS:
Device: repetitive transcranial stimulation (rTMS) — Repetitive TMS will be administered using a MAGSTIM rapid magnetic stimulator (Magstim Company, Ltd., Whitland, U.K.) and a 70-mm figure-eight shaped coils.
  In monolateral treatment in right DLPFC, three 140-second trains will be applied at 1 Hz and at 110% of RMT. There is a 30 seconds intertrain interval (total of 420 stimuli per session). In sequential treatment, the stimulation will be applied in the first to the right and then to the left dorsolateral prefrontal cortex. In right DLPFC will be applied three 140-second trains at 1 Hz and at 110% of RMT. There will be a 30 seconds intertrain interval (total of 420 stimuli per session). In left DLPFC will be applied twenty 5-second trains were applied at 10 Hz and at 100% of RMT. There will be a 25-second intertrain interval (total of 1000 stimuli per session). Patients will be treated from Monday to Friday, for a total of 15 days.
  Arms: 1
Device: unilateral stimulation — Patients will be treated from Monday to Friday, for a total of 15 days in the same timeframe of the active group right sided low frequency stimulation
  Arms: 2

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) has been recently FDA approved for the treatment of resistant depression. No accordance exists on which are the involved mechanisms of action and on which stimulation parameters, frequency and side are optimal.

DETAILED DESCRIPTION:
To compare these different procedures we study patients with unipolar recurrent resistant major depressive disorder in a double-blind, controlled trial randomized to either sequential bilaterally on the right and left dorsolateral prefrontal cortex (DLPFC) or monolaterally on the right DLPFC. Patients will be randomized to receive sequentially low-frequency rTMS at 1 Hz to the right DLPFC and high-frequency rTMS at 10 Hz rTMS to the left DLPFC, or to receive low-frequency rTMS at 1 Hz to the right DLPFC. Significant antidepressant effect as expressed by a reduction of Hamilton Depression Scale score will be recorded in both the groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual-IV criteria for Depressive Major Episode Hamilton Rating Scale for Depression -28 (Ham-D)score ≥ 18
* Failure to respond to a minimum of two courses of antidepressant medications for at least 6 weeks

Exclusion Criteria:

* Any comorbid axis I disorder (except simple and social phobia)
* Any other significant medical, particularly neurologic, illnesses (seizures, head trauma and brain lesions)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAM-D) | at baseline and 3rd week

SECONDARY OUTCOMES:
Clinical Global Impression Scale (CGI) | baseline and 3rd week

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Pallanti, md, Principal Investigator — Istituto di Neuroscienze
Locations (1):
- Institute of Neuroscience, Florence, Italy

REFERENCES:
- [Derived] Pallanti S, Bernardi S, Di Rollo A, Antonini S, Quercioli L. Unilateral low frequency versus sequential bilateral repetitive transcranial magnetic stimulation: is simpler better for treatment of resistant depression? Neuroscience. 2010 May 5;167(2):323-8. doi: 10.1016/j.neuroscience.2010.01.063. Epub 2010 Feb 9. PMID 20144692